CLINICAL TRIAL: NCT06136598
Title: A Phase 1 Clinical Study to Investigate the Safety and Pharmacokinetics of MK-5684 in China Participants With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of Opevesostat (MK-5684) in China Participants With Metastatic Castration-Resistant Prostate Cancer (mCRPC) (MK-5684-001)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5684-001; MK-5684-001 (Other: MSD)
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Prostatic Neoplasms; Metastatic Castration-Resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dexamethasone; dexamethasone acetate; Fludrocortisone; fludrocortisone acetate; Hydrocortisone; hydrocortisone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Opevesostat (Experimental): Participants will receive opevesostat by oral tablets twice daily plus dexamethasone and fludrocortisone by oral tablets once daily continuously until unacceptable toxicity or documented progression. Hydrocortisone will also be provided to participants for use as rescue medication.
  Interventions: Drug: Opevesostat; Drug: Dexamethasone; Drug: Fludrocortisone; Drug: Hydrocortisone

INTERVENTIONS:
Drug: Opevesostat — Tablets to be taken orally.
  Other Names: MK-5684
Drug: Dexamethasone — Tablets to be taken orally
  Other Names: Dexamethasone acetate
Drug: Fludrocortisone — Tablets to be taken orally.
  Other Names: Fludrocortisone acetate
Drug: Hydrocortisone — Tablet to be taken orally as a rescue medication.
  Other Names: Hydrocortisone acetate

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerability of opevesostat in the treatment of male Chinese participants with metastatic castration-resistant prostate cancer (mCRPC) and to characterize the pharmacokinetic profile of opevesostat. There are no formal hypotheses to be tested in this study.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has histologically or cytologically confirmed adenocarcinoma of the prostate without small cell histology.
* Has prostate cancer while receiving androgen deprivation therapy (ADT), or post-bilateral orchiectomy, within 6 months before screening.
* Has evidence of progression >4 weeks since last flutamide treatment or >6 weeks since last bicalutamide or nilutamide treatment.
* Has evidence of metastatic disease documented by either bone lesions on bone scan and/or soft tissue shown by CT/MRI.
* Has disease that progressed during or after treatment with at least 1 line of next-generation hormonal agents (NHAs) for hormone-sensitive prostate cancer (HSPC) or castration-resistant prostate cancer (CRPC) for at least 8 weeks (at least 14 weeks for participants with bone progression).
* Has received at least 1 line of taxane-based chemotherapy for HSPC or CRPC and have had progressed disease during or on treatment, or refused or ineligible to receive chemotherapy.
* Has a life expectancy of >3 months.

Exclusion Criteria:

* Has history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 3 years.
* Has presence of gastrointestinal condition, e.g. malabsorption, that might affect the adsorption of study intervention.
* Has a history of pituitary dysfunction.
* Has poorly controlled diabetes mellitus.
* Has active or unstable cardio/cerebro-vascular disease, including thromboembolic events.
* Has undergone major surgery, including local prostate intervention (except prostate biopsy), within 4 weeks of the date of allocation.
* Has received an anticancer monoclonal antibody (mAb) within 4 weeks of allocation, or has not recovered from adverse events (AEs) due to mAbs administered more than 4 weeks before the date of allocation.
* Received prior systemic anticancer therapy including investigational agents within 4 weeks before the date of allocation.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any form of immunosuppressive therapy within 7 days prior to the start of study intervention.
* Has a known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years.
* Has a history of or current human immunodeficiency virus (HIV) infection.
* Has a concurrent Hepatitis B or Hepatitis C virus infection.
* Has a history of allogenic tissue or solid organ transplant.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2027-03-14 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 20 months
  An AE is defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product and does not imply any judgment about causality.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 20 months
  An AE is defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product and does not imply any judgment about causality.
Maximum Plasma Concentration (Cmax) of opevesostat | Day 1 and Day 8: predose and 0.5, 1, 2, 3, 4, 6, 9, and 12 hours postdose, Day 29, Day 57, and Day 89: pre-dose
  Blood samples will be collected at pre-specified timepoints to determine the Cmax of opevesostat.
Time to Maximum Plasma Concentration (Tmax) of opevesostat | Day 1 and Day 8: predose and 0.5, 1, 2, 3, 4, 6, 9, and 12 hours postdose, Day 29, Day 57, and Day 89: pre-dose
  Blood samples will be collected at pre-specified timepoints to determine the Tmax of opevesostat.
Area Under the Curve from Time 0 to 12 hours postdose (AUC0-12) of opevesostat | Day 1 and Day 8: predose and 0.5, 1, 2, 3, 4, 6, 9, and 12 hours postdose, Day 29, Day 57, and Day 89: pre-dose
  Blood samples will be collected at pre-specified timepoints to determine the AUC0-12 of opevesostat.
Apparent Volume of Distribution (Vz/F) of opevesostat | Day 1 and Day 8: predose and 0.5, 1, 2, 3, 4, 6, 9, and 12 hours postdose, Day 29, Day 57, and Day 89: pre-dose
  Blood samples will be collected at pre-specified timepoints to determine the Vz/F of opevesostat.
Oral Clearance (CL/F) of opevesostat | Day 1 and Day 8: predose and 0.5, 1, 2, 3, 4, 6, 9, and 12 hours postdose, Day 29, Day 57, and Day 89: pre-dose
  Blood samples will be collected at pre-specified timepoints to determine the CL/F of opevesostat.
Half-Life (t1/2) of opevesostat | Day 1 and Day 8: predose and 0.5, 1, 2, 3, 4, 6, 9, and 12 hours postdose, Day 29, Day 57, and Day 89: pre-dose
  Blood samples will be collected at pre-specified timepoints to determine the t1/2 of opevesostat.

SECONDARY OUTCOMES:
Prostate-specific Antigen (PSA) Response Rate | Up to approximately 37 months
  The PSA response rate is defined as the percentage of participants in the analysis population with a reduction in PSA level of ≥50% measured twice ≥3 weeks apart.
Radiographic Progression-free Survival (rPFS) Per Prostate Cancer Working Group (PCWG)-modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 37 months
  rPFS is defined as the time from first dose of study intervention to radiographic progression per PCWG-modified RECIST 1.1 as assessed by the investigator OR death due to any cause, whichever occurs first.
Objective Response Rate (ORR) Per PCWG-modified RECIST 1.1 | Up to approximately 37 months
  ORR is defined as the percentage of participants who have a best overall response of either confirmed Complete Response (CR: disappearance of all target lesions) or a confirmed Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per PCWG-modified RECIST 1.1 as assessed by the investigator.
Duration of Response (DOR) Per PCWG-modified RECIST 1.1 | Up to approximately 37 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per PCWG-modified RECIST 1.1, DOR is defined as the time from first documented evidence of confirmed CR or PR until disease progression or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 37 months
  OS is defined as time from first dose of study intervention to death due to any cause.
Blood Concentrations of Steroids | At designated timepoints (up to approximately 37 months)
  Blood samples collected at multiple timepoints after the administration of opevesostat will be used to determine the blood concentrations of steroids.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (3):
- China (3):
  - Peking University First Hospital-Urology ( Site 0001), Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center-Neurosurgery department ( Site 0003), Guangzhou, Guangdong
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 0002), Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com